CLINICAL TRIAL: NCT01180881
Title: Neurobehavioral Functioning and Utilization of Special Education Services in Pediatric Brain and CNS Tumor Patients After Proton Radiation Treatment: A Longitudinal Study
Brief Title: Neurobehavioral Functioning in Pediatric Brain Tumor Patients After Proton Beam Radiation Treatment
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Margaret Pulsifer, Neuropsychologist, Massachusetts General Hospital
Other Study IDs: 2009A058394
Record Dates: First submitted 2010-08-11; First posted 2010-08-12 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Brain Tumor; Central Nervous System Neoplasms
Keywords: Proton Radiation; CNS tumors; Brain Tumors; Neurobehavioral functioning
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Proton Radiation Patients at MGH: Pediatric brain and central nervous system (CNS) tumor patients treated with proton beam radiation therapy

SUMMARY:
The aim of this study is to follow up with all of the pediatric brain tumor patients who received proton beam radiation therapy at Massachusetts General Hospital (MGH) for which there is baseline neuropsychological testing in order to measure changes, if any, in neurobehavioral functioning (executive skills, emotional/behavioral functioning, and adaptive abilities) and their use of special education services at one year or more post-treatment. The investigators will also correlate neurobehavioral data with pertinent clinical information. Participation will be maximized through the use of mail-in, parental- and self-report questionnaires.

DETAILED DESCRIPTION:
The purpose of this study is to longitudinally examine neurobehavioral functioning outcomes and use of special education services in brain tumor and CNS tumor patients treated with proton radiation at MGH. Furthermore, we seek to correlate neurobehavioral data with pertinent clinical information. We anticipate better neurobehavioral functioning to be associated with use of protons (vs. photons, as reported in the literature). We also anticipate the need and utilization of special education services to be lower in brain and CNS tumor patients treated with protons (vs. photons, as reported in the literature). Lastly, we anticipate greater neurobehavioral deficits in patients whose proton radiation treatment involved the craniospinal axis compared to those who received proton radiation to the involved field.

ELIGIBILITY:
Inclusion Criteria:

1. Children diagnosed with brain or CNS tumors and treated with proton radiation therapy at the MGH Francis H. Burr Proton Center since September 2002
2. Patients received baseline neurocognitive testing at MGH
3. Patients ≤25 years at the time of diagnosis
4. Tumor location in the brain or CNS
5. Radiation treatment consisted of only proton radiotherapy
6. No prior radiation exposure or chemotherapy

Exclusion Criteria:

1. Patients receiving treatment with palliative intent
2. Patients who do not wish to participate
3. Patient is deceased at ≥1 year follow-up

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients who received proton radiation therapy at MGH
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2009-10; Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Behavior Rating Inventory of Executive Functioning | Approximately one year post proton radiation treatment
  Questionnaire of executive functioning in children and young adults
Behavior Assessment System for Children | Approximately one year following proton radiation treatment
  Questionnaire of behavioral functioning in children and young adults
Scales of Independent Behavior-Revised | Approximately one year following proton beam radiation therapy
  Questionnaire of adaptive skills in children and young adults

CONTACTS AND LOCATIONS:
Overall Officials: Margaret B. Pulsifer, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Grieco JA, Evans CL, Yock TI, Pulsifer MB. Psychosocial and executive functioning late effects in pediatric brain tumor survivors after proton radiation. Childs Nerv Syst. 2024 Nov;40(11):3553-3561. doi: 10.1007/s00381-024-06579-2. Epub 2024 Sep 2. PMID 39222091
- [Derived] Pulsifer MB, Duncanson H, Grieco J, Evans C, Tseretopoulos ID, MacDonald S, Tarbell NJ, Yock TI. Cognitive and Adaptive Outcomes After Proton Radiation for Pediatric Patients With Brain Tumors. Int J Radiat Oncol Biol Phys. 2018 Oct 1;102(2):391-398. doi: 10.1016/j.ijrobp.2018.05.069. Epub 2018 Jun 6. PMID 30108004